CLINICAL TRIAL: NCT01178606
Title: Measurement of Echogenic Area in the Border of the Fetal Ventricles
Status: Withdrawn | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10094-2010CTIL
Record Dates: First submitted 2010-08-08; First posted 2010-08-10 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: echogenic halo around lateral fetal ventricles

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Sonographic coronal section in the lateral fetal ventricles shows echogenic area in the ventricles borders creating an "halo" around the ventricles. Histologically this area correlates to the Stratified transitional field. In this study we would like to measure this area for the purpose of creating a nomogram.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 22-37 GA
* well dated pregnancy
* singleton pregnancy

Exclusion Criteria:

* no first trimester dating
* multifetal pregnancy
* known CNS abnormalities in the fetus
* small for gestational age

Ages: 22 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: pregnant women 22-37GA, singleton normal pregnancy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel